CLINICAL TRIAL: NCT04208698
Title: A Randomized, Double-Blind Placebo-Controlled Scintigraphy Study to Investigate the Effect of CIN-102 on Gastric Emptying and Antral Contractility in Adults With Diabetic Gastroparesis
Brief Title: A Scintigraphy Study in Adults With Diabetic Gastroparesis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was terminated due to the impact of COVID-19 on trial activities.
Sponsor: CinDome Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CIN-102-122
Record Dates: First submitted 2019-12-12; First posted 2019-12-23 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Gastroparesis
MeSH Terms: interventions — CIN-102

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CIN-102 Tablets Dose 1 (Experimental): CIN-102 tablets by mouth twice daily for 14 days
  Interventions: Drug: CIN-102 Dose 1
- Placebo for CIN-102 Dose 1 (Placebo Comparator): Placebo tablets by mouth twice daily for 14 days
  Interventions: Drug: Placebo for CIN-102
- CIN-102 Dose 2 (Experimental): CIN-102 tablets by mouth twice daily for 14 days
  Interventions: Drug: CIN-102 Dose 2
- Placebo for CIN-102 Dose 2 (Placebo Comparator): Placebo tablets by mouth twice daily for 14 days
  Interventions: Drug: Placebo for CIN-102

INTERVENTIONS:
Drug: CIN-102 Dose 1 — Deuterated domperidone (deudomperidone)
  Arms: CIN-102 Tablets Dose 1
Drug: CIN-102 Dose 2 — Deuterated domperidone (deudomperidone)
  Arms: CIN-102 Dose 2
Drug: Placebo for CIN-102 — Placebo
  Arms: Placebo for CIN-102 Dose 1; Placebo for CIN-102 Dose 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled scintigraphy study to investigate the effect of oral CIN-102 on gastric emptying and antral contractility in adults with diabetic gastroparesis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled scintigraphy study to investigate the effect of oral CIN-102 on gastric emptying and antral contractility in adults with diabetic gastroparesis. The population for this study is adult patients 18 to 70 years old with Type 1 or Type 2 diabetes and a diagnosis of diabetic gastroparesis. The study will consist of two cohorts with approximately 15 subjects in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 70 years old, inclusive.
* Type 1 or Type 2 diabetes mellitus, according to American Diabetes Association criteria
* Current diagnosis of diabetic gastroparesis.
* Body Mass Index (BMI) between 18 and 40 kg/m2, inclusive.
* Glycosylated hemoglobin level <11% at Screening.
* Willing to abstain from tobacco or nicotine-containing product use after midnight on the day of the DAS test and throughout the time that gastric emptying is being imaged.
* Willing to abstain from grapefruit, grapefruit products, star fruit, star fruit products, and Seville oranges from 72 hours prior to the Randomization Visit until end of study.

Exclusion Criteria:

* History of, or current, clinically significant arrhythmias as judged by the Investigator, including ventricular tachycardia, ventricular fibrillation, atrial fibrillation, and Torsades de Pointes. Patients with minor forms of ectopy (eg, premature atrial contractions) are not necessarily excluded.
* Clinically significant bradycardia with a resting heart rate under 50 beats per minute, sinus node dysfunction, or heart block.
* Prolonged heart rate-corrected QT interval using Fridericia's formula (QTcF) (QTcF >450 msec for males or QTcF >470 msec for females) based on the average of triplicate ECGs.
* A personal or family history of long QT syndrome, Torsades de pointes, or other complex ventricular arrhythmias or family history of sudden death.
* Evidence (based on Screening or Baseline assessments) or history of clinically significant immunologic, hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies); surgical conditions; cancer (with the exception of basal or squamous cell carcinoma of the skin and cancer that resolved or has been in remission for >5 years prior to the Screening Visit); or any condition that, in the Investigator's opinion, might significantly interfere with the absorption, distribution, metabolism, or excretion of the study drug.
* History of prolactin-releasing pituitary tumor (ie, prolactinoma).
* Allergic to egg or intolerant to gluten.
* History of alcoholism or drug abuse within 2 years prior to dosing as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition.
* Known or suspected gastric outlet obstruction (eg, peptic stricture) or other gastrointestinal mechanical obstruction.
* Known history or current diagnosis of intestinal malabsorption or pancreatic exocrine disease.
* History or presence of any medical condition or psychiatric disease, which, in the opinion of the Investigator, could interfere with the conduct of the study or would put the patient at unacceptable risk.
* Judged by the Investigator, after reviewing medical and psychiatric history, physical examination, and laboratory evaluation, to be unsuitable for any other reason that may either place the patient at increased risk during participation or interfere with the interpretation of the study outcomes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Murphy, MD, MPH, Study Director — CinRx Pharma
Locations (1):
- Research Site, El Paso, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients entered the Screening Period. No patients were randomized to the Study Treatment Period.
Groups:
- Screening Period: Screening Period
Period: Overall Study
Arm/Group | Screening Period | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Started | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two patients entered the Screening Period. No patients were randomized to the Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening Period | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2 | Total
Number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  |  | 0
  Between 18 and 65 years | 2 |  |  |  |  | 2
  >=65 years | 0 |  |  |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  |  |  | 1
  Male | 1 |  |  |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  |  |  | 1
  Not Hispanic or Latino | 1 |  |  |  |  | 1
  Unknown or Not Reported | 0 |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 0 | 0 | 0 | 0 | 2
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Change From Baseline in Gastric Percentage Retention of a Radiolabeled Meal After Dosing CIN-102 in Patients With Diabetic Gastroparesis.
Time Frame: Baseline to Day 14
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: To Evaluate the Incidence of Treatment-emergent Adverse Effects as Measured by Safety Laboratory Data and Patient Reported Events.
Time Frame: Screening to Day 20
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: To Assess the Effect of CIN-102 on Antral Contractility as Measured by Dynamic Antral Scintigraphy (DAS), a Non-invasive Technique for the Assessment of Post-prandial Gastric Contractions Will be Used to Evaluate Antral Motility.
Time Frame: Baseline to Day 14
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: To Assess the Effect of CIN-102 on Gastric Accommodation to be Evaluated Using Data Captured During the Total-stomach Gastric Emptying Study to Measure Food Retention in the Stomach During the First Two Post-prandial Hours.
Time Frame: Baseline to Day 14
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: To Asses the Change From Baseline in ANMS GCSI-DD Total Scores
Time Frame: Day -14 to 14
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: To Assess the Change From Baseline in ANMS GCSI-DD Subscale Scores
Time Frame: Day -14 to 14
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: To Assess the Change From Baseline in Symptom Severity as Measured by the PAGI-SYM
Time Frame: Baseline to Day 14
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: To Assess the Change in Baseline of the Clinical Grading Assessment Scale
Time Frame: Baseline to Day 14
Population: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately one month.
Description: No patients were randomized to the study treatment period.
Arm/Group | CIN-102 Tablets Dose 1 | Placebo for CIN-102 Dose 1 | CIN-102 Dose 2 | Placebo for CIN-102 Dose 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04208698/Prot_SAP_001.pdf